CLINICAL TRIAL: NCT05608070
Title: Intravenous Oxytocin for Post Operative Pain After Minimally Invasive Hysterectomy: A Randomized Placebo-Controlled Trial
Brief Title: IV Oxytocin for Post Operative Pain After Minimally Invasive Hysterectomy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor declined to fund
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Lauren Peter, Senior Research Compliance Officer, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P000895
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative; Analgesia; Postoperative Pain; Pain, Post Operative; Oxytocin
Keywords: Postoperative pain; Oxytocin; Non-opioid analgesia; Multimodal analgesia; Female; Humans
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be performed by the Investigational Research Pharmacy. The Investigational Research Pharmacy will have the randomization key and prepare medication or placebo. The study medication or placebo in 500 ml bag of labeled as "Oxytocin Study Drug for IV infusion".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Oxytocin (Experimental)
  Interventions: Drug: Oxytocin
- Placebo- NaCl 0.9% (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 30 IU in 500 ml IV at a rate of 5 IU/h (83.33 ml/h). The infusion will be started intra-operative once the uterus is removed and will continue to run until completion of the medication or discharge from PACU criteria are met, whichever occurs first.
  Other Names: Pitocin
  Arms: IV Oxytocin
Drug: Placebo — 0.9% saline infusion at the rate of 83.3 ml/h.
  Other Names: 0.9% NaCl, Saline
  Arms: Placebo- NaCl 0.9%

SUMMARY:
This double-blinded, placebo-control trial clinical trial aims to investigate the effect of IV oxytocin infusion on peri-operative opioid consumption following a minimally invasive hysterectomy under general anesthesia. The patient population will be women scheduled for an elective, minimally invasive hysterectomy at Beth Israel Deaconess Medical Center.

The investigators hypothesize that, compared to a placebo, exposure to intravenous (IV) oxytocin will reduce the amount of opioid consumption for women after a minimally invasive hysterectomy procedure.

DETAILED DESCRIPTION:
* Patients will be recruited for participation in this study while they are in pre-operative holding area before surgery.
* Once the patient is recruited and consented the patient, they will be randomized for either the intervention group (IV oxytocin) or control group (0.9% normal saline).
* In the holding area, a pre-operative pain questionnaire, including the State-Trait Anxiety Inventory (STAI-6) questionnaire and the Daily Pain Catastrophizing Scale (DPCS), will be performed.
* The STAI-6 is a validated, short 6-question form to assess anxiety. It is one of the most frequently used measures of anxiety in applied psychology research and has been used to assess anxiety in perioperative patients and to assess the potential of a patient to have higher postoperative pain and opioid requirements and a greater likelihood to use chronic opioids or develop chronic pain.
* The DPCS is a validated, short questionnaire to assess measure of catastrophizing in the context of actual or anticipated pain. Similar to the STAI-6, it has been shown to predict patients who experience higher postoperative pain and opioid requirements and those with a greater likelihood of using chronic opioids or developing chronic pain.
* Both groups (intervention and control) will be treated pre-operatively with acetaminophen 1000 mg and gabapentin 300 mg orally.
* The Investigational Research Pharmacy will be informed and prepare medication or placebo.
* The primary anesthesiology team receive either the study medication or placebo in 500 ml bag of labeled as "Oxytocin Study Drug for IV infusion".
* A recommended "Intra-Operative Analgesia Management" algorithm will be given to the primary anesthetic team. The recommended algorithm for intra-operative analgesia management will include the following recommendation:
* Fentanyl 100 mcg IV for induction.
* Dexamethasone 8 mg IV after induction but prior to incision.
* Small, titrated doses of Hydromorphone IV boluses (0.2-0.4 mg) during the operation and before emergence according to primary team judgment.
* Ketorolac 30 mg IV at skin closure unless otherwise contraindicated.
* The infusion will be started intra-operative once the uterus is removed and will continue to run until completion of the medication or discharge from PACU criteria are met, whichever occurs first.
* Other aspects of each patient's routine clinical care will continue as per the attending physician under whom the patient is admitted, regardless of treatment arm status.
* The intervention group will be treated with oxytocin 30 IU in 500 ml IV at a rate of 5 IU/h (83.33 ml/h). The control group will be given IV 0.9% saline infusion at the same rate of 83.3 ml/h. The primary care team (anesthesia, surgery and nurses), research team and the patient will all be blinded for the treatment.
* In the PACU, a brief postoperative pain questionnaire will be done, including the Surgical Pain Scales (SPS).
* The SPS is a validated scale that consists of 4 items that measure pain at rest, during normal activities, during work/exercise and quantify the unpleasantness of worst pain. This scale has been validated in a number of different types of postoperative pain, including women after gynecologic surgery.
* Vital signs, NRS pain scores and opioid consumption at PACU will be collected from the patient's medical record.
* Patients whose surgery was converted to open, EBL >500 ml or any other surgical complication that necessitates a hospitalization will be excluded from the trial.
* For secondary outcomes, including total opioid consumption in 24, 48, and 72 hours and pain scores at POD1, 2, and 3, an online survey will be done at POD1, 2, and 3. For patients who do not complete the survey, a phone call from a study staff member will be performed to complete all questions not completed with the online form.

ELIGIBILITY:
Inclusion Criteria:

* Women the age of 18-65 years old undergoing elective, minimally invasive hysterectomy under general anesthesia

Exclusion Criteria:

* American Society of Anesthesiology (ASA) Physical Status Classification System Score of 4 or greater
* Additional surgical components including but not limited to: minor laparotomy, omentectomy, cystectomy, and lymph node dissection.
* Allergies to any study medication: acetaminophen, ketorolac, hydromorphone, oxycodone, fentanyl, gabapentin, pregabalin.
* Epidural/Regional anesthesia used for intra-operative or post-operative pain.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Total opioids consumption | 3 days
  Average Opioid Oral Morphine Milligram Equivalent (MME) during intra-operative and post-operative period

SECONDARY OUTCOMES:
Post Operative Pain scores | 2 days
  11-point (0-10) pain scores on Numerical Rating Scale (NRS) in Post Anesthesia Care Unit (PACU), Post-Operative Day (POD) 0 and POD1.
Anxiety score | 3 days
  State-Trait Anxiety Inventory (STAI-6)
Quality of Recovery Score | 3 days
  Postoperative Quality of Recovery Score (QoR-15)
Catastrophizing Scale | 3 days
  Daily Pain Catastrophizing Scale (DPCS)
Patient-rated Satisfaction | 1 day
  11-point (0-10) patient satisfaction scores on Numerical Rating Scale (NRS) in PACU and POD0

CONTACTS AND LOCATIONS:
Overall Officials: John J. Kowalczyk, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Shiri Savir, MD MPH, Study Director — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soffin EM, Lee BH, Kumar KK, Wu CL. The prescription opioid crisis: role of the anaesthesiologist in reducing opioid use and misuse. Br J Anaesth. 2019 Jun;122(6):e198-e208. doi: 10.1016/j.bja.2018.11.019. Epub 2018 Dec 28. PMID 30915988
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Bae S, Alboog A, Esquivel KS, Abbasi A, Zhou J, Chui J. Efficacy of perioperative pharmacological and regional pain interventions in adult spine surgery: a network meta-analysis and systematic review of randomised controlled trials. Br J Anaesth. 2022 Jan;128(1):98-117. doi: 10.1016/j.bja.2021.08.034. Epub 2021 Nov 10. PMID 34774296
- [Background] Lundeberg T, Uvnas-Moberg K, Agren G, Bruzelius G. Anti-nociceptive effects of oxytocin in rats and mice. Neurosci Lett. 1994 Mar 28;170(1):153-7. doi: 10.1016/0304-3940(94)90262-3. PMID 8041495
- [Background] Biurrun Manresa JA, Schliessbach J, Vuilleumier PH, Muller M, Musshoff F, Stamer U, Stuber F, Arendt-Nielsen L, Curatolo M. Anti-nociceptive effects of oxytocin receptor modulation in healthy volunteers-A randomized, double-blinded, placebo-controlled study. Eur J Pain. 2021 Sep;25(8):1723-1738. doi: 10.1002/ejp.1781. Epub 2021 May 3. PMID 33884702
- [Background] Gimpl G, Fahrenholz F. The oxytocin receptor system: structure, function, and regulation. Physiol Rev. 2001 Apr;81(2):629-83. doi: 10.1152/physrev.2001.81.2.629. PMID 11274341
- [Background] Baribeau DA, Anagnostou E. Oxytocin and vasopressin: linking pituitary neuropeptides and their receptors to social neurocircuits. Front Neurosci. 2015 Sep 24;9:335. doi: 10.3389/fnins.2015.00335. eCollection 2015. PMID 26441508
- [Background] Miranda-Cardenas Y, Rojas-Piloni G, Martinez-Lorenzana G, Rodriguez-Jimenez J, Lopez-Hidalgo M, Freund-Mercier MJ, Condes-Lara M. Oxytocin and electrical stimulation of the paraventricular hypothalamic nucleus produce antinociceptive effects that are reversed by an oxytocin antagonist. Pain. 2006 May;122(1-2):182-9. doi: 10.1016/j.pain.2006.01.029. Epub 2006 Mar 9. PMID 16527400
- [Background] Madrazo I, Franco-Bourland RE, Leon-Meza VM, Mena I. Intraventricular somatostatin-14, arginine vasopressin, and oxytocin: analgesic effect in a patient with intractable cancer pain. Appl Neurophysiol. 1987;50(1-6):427-31. doi: 10.1159/000100753. PMID 2897190
- [Background] Yang J. Intrathecal administration of oxytocin induces analgesia in low back pain involving the endogenous opiate peptide system. Spine (Phila Pa 1976). 1994 Apr 15;19(8):867-71. doi: 10.1097/00007632-199404150-00001. PMID 8009342